CLINICAL TRIAL: NCT00131586
Title: Cisplatin, Carboplatin, and Oxaliplatin Interactions With Plasma Proteins
Status: Terminated | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: SP-11-0033/ethics 17173
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2012-04

CONDITIONS: Lung Cancer; Colorectal Cancer
Keywords: platinum analogues; cisplatin, carboplatin, oxaliplatin; proteomics; hemoglobin
MeSH Terms: conditions — Lung Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cisplatin is a widely used anti-tumor agent for the treatment of testicular and ovarian cancers. Carboplatin is used extensively for small cell, non small cell lung cancer and ovarian cancer. Oxaliplatin has recently been approved in the United States (US) for treatment of colorectal cancer. A large portion (in the range of 65% to 98%) of cisplatin in the blood plasma was bound to protein within a day after intravenous administration. The binding of cisplatin and other analogues to proteins and enzymes is generally believed to be the cause of several severe side effects such as ototoxicity and nephrotoxicity. The interactions between platinum based chemotherapy drugs and proteins is proposed to play important roles in both drug activity and toxicity. Therefore, a better understanding of the molecular mechanism of platinum-protein interactions may have an impact on optimization of strategies for treatment. The objective is to develop novel approaches and techniques to provide detailed mechanistic, kinetic and high-resolution structural information on the binding of platinum analogues to blood proteins, and to improve treatment efficacy and reduce side effects.

DETAILED DESCRIPTION:
Cisplatin, cis-[Pt(NH3)2Cl2], is a widely used antitumor agent for the treatment of testicular and ovarian cancers. Carboplatin is used extensively for small cell, non small cell lung cancer and ovarian cancer. Oxaliplatin has recently been approved in the US for treatment of colorectal cancer. All of these analogues are administered by intravenous injection, and within one day, 65-98% of the platinum in the blood plasma is bound to protein. Binding of cisplatin to proteins reduces urinary excretion of platinum, and causes deposition of platinum in tissues. Binding of cisplatin to proteins and enzymes is generally believed to be the cause of several severe side effects exhibited by these drugs, especially ototoxicity and nephrotoxicity.

Despite numerous studies of platinum-protein binding in the last few decades, the roles of platinum-protein adducts in drug action, and in toxicity of these drugs are not known. Although cisplatin-protein adducts are widely believed to cause the drug's side effects, there are also claims that platinum-protein adducts are important for the drug's activity. Therefore, a better understanding of the molecular mechanism of platinum-protein interactions may have an impact on the optimization of strategies for platinum treatment. It is important to understand basic principles that govern formation and reactivity of platinum-protein adducts because these adducts may be important in defining the therapeutic profile of these drugs. In this quest, the first goal is to develop a reliable technique for these studies. To date, ultraviolet/visible (UV-Vis), fourier transform infrared (FT-IR), and nuclear magnetic resonance (NMR) studies of cisplatin-protein interactions have provided only low-resolution information on the mechanism of the binding or on the nature of the adducts. The researchers propose to investigate the role of platinum-protein adducts in the mechanisms of the drug action and their contributions towards the toxicity of these drug. The short-term objective is to investigate platinum interaction with serum proteins using both nanoelectrospray mass spectrometry (nanoESI-MS) and a combination of size exclusion high performance liquid chromatography with inductively coupled plasma mass spectrometry (HPLC/ICP-MS). The long-term objective of this research is to develop biomarkers based on platinum-protein adducts for clinical monitoring.

Initially, metallothionein and human hemoglobin were used as model proteins to develop nESI/MS and HPLC/ICP-MS techniques for studying cisplatin-protein interactions in vitro. The researchers have demonstrated that the combination of size exclusion HPLC/ICP-MS and nanoESI/MS provided new information on the adduct formation and potential reaction mechanism. The size exclusion HPLC with ICP-MS enables monitoring of cisplatin-protein binding under physiological conditions. Nanospray tandem MS offers information on formation of specific complexes and on characteristics of binding. This information is useful for a better understanding of drug toxicity and treatment resistance. The information on platinum-protein interactions allows us to evaluate the utility of both nanoESI/MS and size exclusion HPLC/ICP-MS techniques in providing mechanistic, kinetic and structural information on the binding of platinum to other proteins. The methodology will be further validated by studying the platinum-blood protein adducts in cancer patients undergoing chemotherapeutic treatments. The correlation between the levels of platinum-protein adducts and clinical outcomes will be studied.

The successful completion of this research program should provide the researchers with a better understanding of mechanisms of the drug action and toxicity. This knowledge will be of great importance in clinical monitoring of cancer patients to assist doctors to improve cancer chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* To have lung or colorectal cancer and be treated with either oxaliplatin, carboplatin or cisplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2003-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sawyer, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada